CLINICAL TRIAL: NCT00058747
Title: Phase II Exploratory Study Of AG-858 Plus Gleevec™ In Patients With Chronic Myelogenous Leukemia (CML) In Chronic Phase Who Are Cytogenetically Positive After Treatment With Gleevec™
Brief Title: AG-858 in Patients Who Are Cytogenetically Positive After Treatment With Gleevec™
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision of the sponsor
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-300-01; NCT00070395 (obsolete NCT alias)
Record Dates: First submitted 2003-04-11; First posted 2003-04-15 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Leukemia, Myeloid, Chronic
Keywords: Granulocytic Leukemia, Chronic; Leukemia, Granulocytic, Chronic; Leukemia, Myelocytic, Chronic; Leukemia, Myelogenous, Chronic; Myelocytic Leukemia, Chronic; Myelogenous Leukemia, Chronic; Myeloid Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

INTERVENTIONS:
Drug: Autologous HSP-70 Protein-Peptide Complex (AG-858) Plus Gleevec™.

SUMMARY:
This is a Phase II, exploratory, open-label study of the investigational product AG-858, in patients who are cytogenetically positive after treatment with Gleevec.

The trial will consist of three independent Phase II evaluations of patient groups according to their cytogenetic status as defined in the eligibility criteria (Eligibility Criteria 4a, 4b, and 4c).

DETAILED DESCRIPTION:
The goals of this study are to determine the following:

* To estimate the proportion of patients with a complete cytogenetic response (CCR) within each patient group
* To estimate the proportion of patients with a substantial molecular response (SMR) within each patient group
* To evaluate the frequency and severity of adverse events.
* To assess the feasibility of AG-858 production.

ELIGIBILITY:
Inclusion Criteria:

* Must be Philadelphia chromosome positive chronic myelogenous leukemia in first chronic phase
* Must have a complete hematologic response
* Must have received Gleevec™, IFN-α, cytarabine, busulfan, hydroxyurea, Homoharringtonine (HHT) or any combination thereof as long as the combination has been discontinued and the dosing of Gleevec™ has been stable for 6 months or greater
* Must have one of the following cytogenetic statuses:

(A) Less than a CCR after receiving Gleevec™ for at least one year at a minimum dose of 400 mg/day. A stable dose of Gleevec™ must have been maintained for the last six months prior to eligibility testing OR (B) Stable cytogenetic status without CCR (no cytogenic response or progression) in three consecutive determinations over six months while on a stable dose of Gleevec™ (at a minimum of 400mg/day) for at least 6 months OR (C) Cytogenetic progression while on a stable dose of Gleevec™ (at a minimum dose of 400mg/day)for at least 2 consecutive evaluations at least one month apart

* ECOG performance score of 0 or 1
* Must be at least 18 years old
* Not pregnant or breastfeeding and agree to use contraception during the course of the study
* No prior allogeneic bone marrow transplant or be candidates for curative BMT
* No immunodeficiency or other serious illness
* No current use of immunosuppressive medications
* No other cancer within the last five years, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri or basal or squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-03; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (11):
  - Birmingham, Alabama
  - La Jolla, California
  - Los Angeles, California
  - Denver, Colorado
  - Farmington, Connecticut
  - Chicago, Illinois
  - Boston, Massachusetts
  - St Louis, Missouri
  - New York, New York
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
- United Kingdom (2):
  - Liverpool
  - London

REFERENCES:
- See also: For more information regarding Gleevec™, please visit Novartis' website — http://www.novartis.com